CLINICAL TRIAL: NCT06695026
Title: A Phase 1b/2a, Open-label, Multicenter, Randomized, Dose Escalation Study Evaluating the Safety, Tolerability and Efficacy of RZ-001 in Combination With Valganciclovir and Atezolizumab/Bevacizumab in Subjects With Hepatocellular Carcinoma
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of RZ-001 in Combination With Valganciclovir (VGCV) and Atezolizumab/Bevacizumab in Subjects With Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rznomics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RZ-001-102
Record Dates: First submitted 2024-11-06; First posted 2024-11-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 (Experimental): o Interventions:
  Drug: RZ-001 Dose 1
  Interventions: Drug: RZ-001 Dose 1
- Cohort 2 (Experimental): o Interventions: Drug: RZ-001 Dose 2
  Interventions: Drug: RZ-001 Dose 2
- Cohort 3 (Experimental): o Interventions: Drug: RZ-001 Dose 3
  Interventions: Drug: RZ-001 Dose 3

INTERVENTIONS:
Drug: RZ-001 Dose 1 — RZ-001 Dose 1 and VGCV, Atezolizumab/Bevacizumab
  Arms: Cohort 1
Drug: RZ-001 Dose 2 — RZ-001 Dose 2 and VGCV, Atezolizumab/Bevacizumab
  Arms: Cohort 2
Drug: RZ-001 Dose 3 — RZ-001 Dose 3 and VGCV, Atezolizumab/Bevacizumab
  Arms: Cohort 3

SUMMARY:
This study is to evaluate the safety, tolerability, efficacy and immunogenicity of RZ-001 in combination with Valganciclovir (VGCV) and Atezolizumab/Bevacizumab when given to subjects with human telomerase reverse transcriptase (hTERT)-positive HCC.

DETAILED DESCRIPTION:
15 subjects will be enrolled in each of the 3 cohorts. Once enrollment of the first 3 of 15 subjects is completed, Safety and Efficacy Review Committee (SERC) meeting involving the study Investigators and the Sponsor's clinical study team will be held after Day 43 (Week 6) visit of the third subject enrolled. After the data from enrolled subjects is reviewed in the meeting, dose escalation to the next dose will be determined, based on the number of subjects experiencing dose-limiting toxicity (DLT).

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females
* Hepatocellular carcinoma diagnosis (BCLC stage B or C)
* hTERT positive expression confirmed during the screening period
* ECOG score of 0 or 1
* Child-Pugh score of A
* Life expectancy >= 3 months

Exclusion Criteria:

* Moderate or severe ascites
* History of hepatic encephalopathy
* Carcinomas other than HCC
* Current or history of HIV positive
* Not suitable for inclusion judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) as graded by NCI CTCAE | Screening visit, up to 2 years
Assessment of tumor response of target lesion where RZ-001 is administered based on the RECIST v1.1 and HCC mRECIST | Screening visit, every 2 cycles (each cycle is 3 weeks, 6 weeks) until week 54 & every 3 cycles (each cycle is 3 weeks, 9 weeks) after week 54, up to 2 years
Overall response rate based on RECIST v1.1 and HCC mRECIST | Screening visit, every 2 cycles (each cycle is 3 weeks, 6 weeks) until week 54 & every 3 cycles (each cycle is 3 weeks, 9 weeks) after week 54, up to 2 years

SECONDARY OUTCOMES:
Assessment of tumor response of non-target lesions, besides the target lesion where RZ-001 is administered based on the RECIST v1.1 and HCC mRECIST | Screening visit, every 2 cycles (each cycle is 3 weeks, 6 weeks) until week 54 & every 3 cycles (each cycle is 3 weeks, 9 weeks) after week 54, up to 2 years
Progression-free survival (PFS) | Screening visit, every 2 cycles (each cycle is 3 weeks, 6 weeks) until week 54 & every 3 cycles (each cycle is 3 weeks, 9 weeks) after week 54, up to 2 years
Overall survival (OS) | Screening visit, every 2 cycles (each cycle is 3 weeks, 6 weeks) until week 54 & every 3 cycles (each cycle is 3 weeks, 9 weeks) after week 54, up to 2 years
Duration of response (DOR) | Screening visit, every 2 cycles (each cycle is 3 weeks, 6 weeks) until week 54 & every 3 cycles (each cycle is 3 weeks, 9 weeks) after week 54, up to 2 years

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Pusan National University Yangsan Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No